CLINICAL TRIAL: NCT04441294
Title: The Evaluation of Achieving Condom Empowerment (ACE)-Plus in New York City
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Philliber Research & Evaluation (Other)
Collaborators: The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott Herrling, Senior Research Associate, Philliber Research & Evaluation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PhiiliberCAI
Record Dates: First submitted 2020-06-15; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Teen Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACE-Plus (Experimental): ACE-Plus is a one-on-one dual-session intervention for males aged 16 to 20 within foster care or preventive services settings which promotes condom use and knowledge of dual methods of contraception. The goal of ACE-Plus is to promote correct and consistent condom use of male latex condoms during penile-vaginal sex and to promote male engagement (e.g., discussion, decision-making) with their female partners in the use of female-centered contraception methods.
  Session one focuses on correct and consistent condom use for purposes of HIV/STD prevention including information and activities that address teen pregnancy prevention. Session two, which occurs within 10 to 14 days of the first session, promotes dual-method contraceptive use. Both sessions are one hour.
  Interventions: Behavioral: ACE-Plus
- On Track (No Intervention): On Track was the alternative program provided to males randomly assigned to the control group. On Track seeks to assist participants in identifying their aptitudes and preferences regarding their careers and their values associated with employment, and to provide tools to prepare them for the work setting and future job interviews. Participants learn how to identify attitudes, values, preferences, and challenges surrounding a career path, receive an understanding of the documents required for employment, and develop an initial employment strategy and action plan. Trained foster care agency staff deliver the curriculum to participating youth in two one-on-one sessions at agencies. Each session is one hour in length. Session two occurs 10 to 14 days after session one.

INTERVENTIONS:
Behavioral: ACE-Plus
  Arms: ACE-Plus

SUMMARY:
To test a new curriculum - the ACE-Plus curriculum - a two-session program that teaches males in foster care and/or preventive services about correct and consistent condom use as well as engagement with female partners to obtain and use contraception.

DETAILED DESCRIPTION:
ACE-Plus is a one-on-one dual-session intervention for males aged 16 to 20 within foster care or preventive services settings which promotes condom use and knowledge of dual methods of contraception. The goal of ACE-Plus is to promote correct and consistent condom use of male latex condoms during penile-vaginal sex and to promote male engagement (e.g., discussion, decision-making) with their female partners in the use of female-centered contraception methods.

Over 200 males aged 16 to 20 were recruited into this study (called My Plan) by 9 foster care agencies in New York City from June 2016 through November 2019. The foster care agencies were selected by Cicatelli Associates, Inc. in New York City, a non-profit organization which oversaw the implementation of the study. These agencies represent a convenience sample which agreed to participate and deliver either the treatment condition (Ace-Plus) or a benign control condition (On Track). Agency staff received a five-day training regarding the implementation of both programs prior to youth engagement and also received additional refresher trainings and technical assistance as needed.

Agency staff screened potential study youth to ascertain eligibility. To be eligible for inclusion in this study, interested youth must have been born with a penis, been aged 16 to 20, have had vaginal intercourse at least once, and could not be currently participating in any other teen pregnancy prevention program. Targeted youth were either in foster care or preventive services. Screening occurred until 238 males were enrolled and completed a baseline assessment.

After youth met the screening criteria and agreed to participate, agency staff obtained written parental consent (from biological parents) and youth assent for each male age 16 or 17 to participate in the study. Participants who were 18 to 20 years old provided their own written consent. Staff obtained written consent for freed minors from the Commissioner of Administration for Children's Services in New York City. Consent forms included consent for both program participation and participation in the evaluation. Both English and Spanish consent forms were utilized.

All study procedures were approved by three Institutional Review Boards: the Administration for Children's Services in New York City, the New York State Office of Children and Family Services, and Advarra® - a national IRB.

After a youth was deemed eligible to participate and had proper written consent and assent, he completed a baseline survey via SurveyMonkey at the foster care agency. Randomization occurred at the time of the final question on the baseline survey, which prompted the youth to draw a chip from a bag. The color of the chip determined group assignment. Trained agency staff oversaw this process to ensure accuracy.

Assigned youth then received the first of two one-hour sessions, with the second session occurring 10 to 14 days after the first. This is an intent-to-treat randomized controlled trial which includes all randomized youth regardless of dosage.

Follow-up assessments were completed 3- and 9-months after the end of session two. The evaluators followed-up with participants via email, text, phone, and regular mail to have them complete the 3- and 9-month follow-up surveys. A $50 stipend was provided to youth at the end of session two, for completion of the 3-month follow-up survey, and for completion of the 9-month follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

1. Youth must have been born with a penis
2. Youth must be aged 16 to 20
3. Youth must have had vaginal intercourse at least once
4. Youth can not be currently participating in any other teen pregnancy prevention program
5. Youth must be in foster care or preventive services

Exclusion Criteria:

1. Lack of consent.

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 238 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Condom use in the past 3 months | 3-month follow-up
  The primary outcome of interest focused on condom use in the past three months at 3-month follow-up. On all surveys, youth were asked the following question:
  In the past three months, how many times have you had vaginal sex without using a condom?
Condom use in the past 3 months | 9-month follow-up
  The primary outcome of interest focused on condom use in the past three months at 9-month follow-up. On all surveys, youth were asked the following question:
  In the past three months, how many times have you had vaginal sex without using a condom?

SECONDARY OUTCOMES:
Use of hormonal birth control methods (birth control pills, shot, patch, ring, IUD, or implants) while having vaginal sex during the past 3 months. | 3-month follow-up
  The first secondary research question focused on use of hormonal birth control methods (birth control pills, shot, patch, ring, IUD, or implants) while having vaginal sex during the past three months. On all surveys, youth were asked the following question:
  In the past three months, how many times have you had vaginal sex without using an effective method of birth control (birth control pills, shot, patch, ring, IUD, or implants)?
Use of birth control by female partner(s) | 3-month follow-up
  The second secondary research question involved use of birth control by female partner(s). On all surveys, youth were asked:
  In the past 3 months, how often do you think your female sex partner(s) were using birth control?
Obtaining birth control | 3-month follow-up
  The third secondary research question involved obtaining birth control with sexual partner(s). On all surveys, youth were asked:
  In the past 3 months, have you been to a clinic or doctor with your sexual partner(s) to obtain birth control?
Communication with sexual partner(s) about birth control | 3-month follow-up
  The fourth secondary research question involved communication with sexual partner(s) about birth control. On all surveys, youth were asked:
  In the past 3 months, how often have you spoken with your sexual partner(s) about the type of birth control they are using?

IPD SHARING:
Plan to Share IPD: No